CLINICAL TRIAL: NCT02543593
Title: Efficacy of Transcranial Direct-Current Stimulation (tDCS) for Provoked Vestibulodynia : a Triple Blind Randomized Controlled Trial
Acronym: PVD/tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mélanie Morin, pht, PhD, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-169
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Provoked Vestibulodynia
Keywords: tDCS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants will receive active transcranial direct-current stimulation (tDCS) for ten 20 minute sessions of 2 mA stimulation over a 2-week period.
  Interventions: Device: Active tDCS or Sham tDCS
- Placebo (Sham Comparator): Participants will receive sham transcranial direct-current stimulation (tDCS) for ten 20 minute sessions of 2 mA stimulation over a 2-week period.
  Interventions: Device: Active tDCS or Sham tDCS

INTERVENTIONS:
Device: Active tDCS or Sham tDCS — tDCS is a painless technique which consists in applying low direct-current through electrodes (one electrode serving as an anode, the other as a cathode) placed on the scalp to target the cerebral cortex. In patients with chronic pain, the anode is commonly placed over the motor cortex (M1) (Valeriani et al., 1999).
  Other Names: neuroConn; Model no: 0008; Serial no:0169

SUMMARY:
Provoked vestibulodynia (PVD) is the most common form of vulvodynia and despite its high prevalence and important sexual, conjugal and psychological deleterious repercussions, effective evidence-based interventions remain limited. For a high proportion of women, significant pain persists despite the currently available treatments. Transcranial direct-current stimulation (tDCS) was shown to be effective in various chronic pain conditions. So far, only one case report study has shown significant pain reduction in women with vulvodynia. The main goal of this randomized controlled trial is to evaluate the efficacy of tDCS in women with PVD compared to sham tDCS. Forty women diagnosed with PVD, by a gynecologist following a standardized protocol will be randomized to either active or sham tDCS for ten 20 minute sessions of 2 mA stimulation over a 2-week period. Outcome measures will be collected at baseline, after treatment and at 3-month follow-up. The primary outcome is pain during intercourse assessed with a numerical rating scale (NRS). Secondary measurements focus on sexual function, vestibular pain sensitivity, psychological distress, treatment satisfaction and Patient Global Impression of Change (PGIC). The investigators expect that active tDCS treatment will significantly reduce pain during intercourse (post-treatment and 3-month follow-up compared to pre-treatment assessment). This trial will provide important information for determining the efficacy of a novel and promising intervention for women with PVD.

ELIGIBILITY:
Inclusion Criteria:

1. Experience moderate to severe pain in at least 90% of attempted sexual intercourse;
2. Experience moderate to severe pain during cotton swab test, in one or more regions of the vestibule (minimum of 5/10 on a subjective numeric scale of pain intensity);
3. Pain limited to the vestibule during vaginal intercourse and during activities exerting pressure on the vestibule (tampon insertion, tight jeans or pants, cycling, horseback riding);
4. Presence of PVD for at least 6 months and diagnosed according to the standardized gynecological examination protocol by one of our staff gynecologists;
5. Have a stable sexual partner with regular sexual activity including penetration.

Exclusion Criteria:

1. Other pelvic pathology associated with pelvic pain (e.g., deep dyspareunia);
2. Chronic pain conditions (e.g. fibromyalgia, low back pain, chronic migraines);
3. Use of medication that can influence the perception of pain (eg analgesic, opioids, antiepileptic, muscle relaxant);
4. Pregnancy for less than one year and breastfeeding;
5. Anterior vulvar or vaginal surgery;
6. Refusal to refrain from other treatments one month prior to first treatment study until the last 3-month follow-up assessment;
7. Important urogynecologic symptoms (urinary or anal incontinence, urinary urgency, pelvic organ prolapse, active urinary tract or vaginal infection or earlier in the last 3 months, etc.);
8. Contraindications to tDCS (e.g. metallic implant in or near the skull, history of epilepsy, pacemaker);
9. Previously received tDCS treatment.

Ages: 17 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pain during intercourse (Numeric rating scale) | Change in the NRS scores from pre- to 2-week post-treatment, and from pre-treatment to 3-month post-treatment
  Pain during intercourse will be assessed using a numeric rating scale (NRS) ranging from 0 to 10, where 0 is no pain at all, and 10 is the worst pain ever. This method for measuring pain has been shown to detect significant treatment effects in women with PVD and demonstrates a significant positive correlation with other pain intensity measures. Pain during intercourse is the main symptom of PVD and the one that most interferes with quality of life, hence the most relevant measure of functional outcome (Bergeron et al., 2008; Bergeron et al., 2001; Morin et al., 2010; Morin et al., 2011).

SECONDARY OUTCOMES:
Pain (McGill-Melzack questionnaire) | Change in the McGill-Melzack scores from pre- to 2-week post-treatment, and from pre-treatment to 3-month post-treatment
  The McGill-Melzack questionnaire allows the assessment of sensory, affective and evaluative components of pain. This world-renowned questionnaire, studied for its validity, reliability and responsiveness to change, is commonly used in RCTs (Bergeron et al., 2001; Melzack, 1975; Davidoff et al., 1987; Hays et al., 1994; Bansal et al., 2009; Moy et al., 2011; Foster et al., 2010).
Vestibular sensitivity (algometer) | Change in the pain threshold and pain tolerance scores from pre- to 2-week post-treatment, and from pre-treatment to 3-month post-treatment
  A gradual pressure (1 to 1000 g) will be applied to three distinct points of the vestibule at the 3, 6 and 9 o'clock positions (Cyr et al., 2014). Each of these pressure points will be applied randomly (e.g. 3,6,9 or 3,9,6 or 6,9,3.). During this procedure, each participant will be asked to indicate when they start to feel pain (pain threshold) and subsequently the maximal pressure that can be tolerated (pain tolerance). Pain intensity is assessed throughout the test using a Computerized Visual analog scale (CoVas). This assessment has shown good reliability and validity (Cyr et al., 2014).
Female Sexual Function Index (FSFI) | Change in the FSFI scores from pre- to 2-week post-treatment, and from pre-treatment to 3-month post-treatment
  The Female Sexual Function Index (FSFI) is a multidimensional measure of sexual function evaluating desire, arousal, lubrication, orgasm, satisfaction and pain. In addition to good psychometric properties (reliability, internal consistency and responsiveness to change (Rosen et al., 2000; Goldfinger et al, 2009), normative data are available for this questionnaire suggesting clinical level of dysfunctions (Wiegel et al., 2005).
Pain Catastrophizing Scale (PCS) | Change in the PCS scores from pre- to 2-week post-treatment, and from pre-treatment to 3-month post-treatment
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (Sullivan, Bishop, & Pivik, 1995), which consists of 13 items measuring exaggerated negative thoughts and feelings about the meaning of pain. Items are scored on a 5-point scale with the end points (0) not at all and (4) all the time. The PCS is a reliable and valid measure that has demonstrated a stable factorial structure across clinical and general populations, including a French population (French et al., 2005; Osman et al., 2000; Sullivan, et al., 1995).
Spielberg State-Trait Anxiety Inventory (IASTA) | Change in the IASTA state and IASTA trait scores from pre- to 2-week post-treatment, and from pre-treatment to 3-month post-treatment
  Anxiety will be assessed using the Spielberger State-Trait Anxiety Inventory (STAI - (Spielberger, Gorsuch, & Lushene, 1970); ASTA - (Gauthier & Bouchard, 1993)). The STAI is a 40-item, well-known and widely used measure of state and trait anxiety that has demonstrated very good psychometric properties (Cronbach's alpha State = .93, Trait = .97) in various clinical and non-clinical samples including pain populations (Gauthier & Bouchard, 1993; Greenberg & Burns, 2003; Rule & Traver, 1983; Tanaka-Masumi & Kameoka, 1986).
Beck Depression Inventory questionnaire (BDI-II) | Change in the BDI scores from pre- to 2-week post-treatment, and from pre-treatment to 3-month post-treatment
  Depression or depression symptoms will be measured with the Beck Depression Inventory-II (BDI-II). The BDI-II is comprised of 21 items, with scores for most items ranging from 0 (low intensity) to 3 (high intensity) (Beck, Steer & Brown, 1996; Beck, Steer & Garvin, 1988). This measure of depression has been validated for use in chronic pain populations (Turner & Romano, 1984).
Pain Anxiety Symptoms Scale (PASS-20) | Change in the PASS-20 scores from pre- to 2-week post-treatment, and from pre-treatment to 3-month post-treatment
  The Pain Anxiety Symptoms Scale (PASS-20), evaluating fear of pain, also shows good psychometric properties (Coons, Hadjistavropoulos & Asmundson, 2004; McCracken & Dhingra, 2002).
Patient's global impression of change (PGIC) | Change in the PGIC scores from 2-week post-treatment to 3-month post-treatment
  Patient self-reported improvement [scale of 0 (completely dissatisfied) to 10 (completely satisfied)] and treatment satisfaction [scale of 0 (worse) to 10 (complete cure)] will be measured at the 2-week post-treatment and 3-month post-treatment structured interview in order to assess the clinical significance of results.
Global Measure of Sexual Satisfaction scale (GMSS) | Change in the GMSS scores from pre- to 2-week post-treatment, and from pre-treatment to 3-month post-treatment
  Sexual satisfaction will be assessed using the Global Measure of Sexual Satisfaction scale, which consists of 5 items assessing global sexual satisfaction. Internal consistency of this scale is high (alpha = 0.90), as is test-retest reliability (r = 0.84) (Lawrance & Byers, 1998).

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Centre hospitalier Universitaire de Sherbroke, Sherbrooke, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Derived] Morin A, Leonard G, Gougeon V, Waddell G, Bureau YA, Girard I, Morin M. Efficacy of transcranial direct-current stimulation (tDCS) in women with provoked vestibulodynia: study protocol for a randomized controlled trial. Trials. 2016 May 14;17(1):243. doi: 10.1186/s13063-016-1366-5. PMID 27179944
- See also: Facebook page — https://www.facebook.com/pages/Laboratoire-de-recherche-en-urogyn%C3%A9cologie/277240805641504?fref=ts
- See also: Laboratory Web page — http://www.lab-urogyn.com/